CLINICAL TRIAL: NCT00235560
Title: Rapamycin in Combination With Low-dose Aracytin in Elderly Acute Myeloid Leukemia Patients. A Study From the Groupe Ouest Est d'étude Des Leucémies Aiguës Myéloïdes (GOELAMS)
Brief Title: Rapamycin in Combination With Low-dose Aracytin in Elderly Acute Myeloid Leukemia Patients
Acronym: LAM-RAPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0402008; GOELAMS; PHRC
Record Dates: First submitted 2005-09-09; First posted 2005-10-10 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Rapamycin; Elderly; Elderly patients not eligible for intensive chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapamycine (Experimental)
  Interventions: Drug: rapamycin

INTERVENTIONS:
Drug: rapamycin — sirolimus
  Other Names: RAPAMUNE

SUMMARY:
These study is designed to evaluate the tolerability and efficacy of sirolimus (rapamycin) in combination with low-dose aracytin in elderly AML.

DETAILED DESCRIPTION:
Evaluate the tolerability and efficacy of sirolimus (rapamycin) in combination with low-dose aracytin

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* de novo or secondary LAM (CML excluded) not elligible for intensive chemotherapy.
* Previously untreated

Exclusion Criteria:

* Renal impairment (serum creatinin >2N)
* Hepatic impairment (TGO ou TGP > 5N), une cholestase (Phosphatases Alcalines or gamma-GT > 5N),bilirubin > 3N

  * Blast crisis CML
  * Acute Promyelocytic Leukemia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
tolerability
bioclinical markers of response

CONTACTS AND LOCATIONS:
Overall Officials: RECHER Christian, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - Service d'Hématologie, CHU, Angers
  - Service d'Hématologie, Hôpital Jean Minjoz, Besançon
  - Service d'Hématologie CHU Purpan, Toulouse

REFERENCES:
- [Background] Recher C, Beyne-Rauzy O, Demur C, Chicanne G, Dos Santos C, Mas VM, Benzaquen D, Laurent G, Huguet F, Payrastre B. Antileukemic activity of rapamycin in acute myeloid leukemia. Blood. 2005 Mar 15;105(6):2527-34. doi: 10.1182/blood-2004-06-2494. Epub 2004 Nov 18. PMID 15550488